CLINICAL TRIAL: NCT00302406
Title: Naturalistic Substitution of Concerta in Adult Subject With ADHD Receiving Immediate Release Methylphenidate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Thomas J. Spencer, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003-P-000038
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate hydrochloride
Drug: OROS methylphenidate hydrochloride (CONCERTA)

SUMMARY:
This is a single-blind study looking at the efficacy and satisfaction of Concerta substitution in adult subjects with ADHD receiving immediate release methylphenidate. Subjects will be administered a maximum dose of 1.3mg/kg/day of either methylphenidate or Concerta. The specific hypotheses of this study are:

Hypothesis 1: ADHD symptomatology in adults with DSM-IV, ADHD will continue to be controlled in patients switched from MPH IR TID to Concerta.

Hypothesis 2: Patient satisfaction will not decrease in patients switched from MPH IR TID to Concerta (ie., all patients will be equally or more satisfied on Concerta as compared with MPH IR TID.

DETAILED DESCRIPTION:
Concerta was specifically developed to replace three times a day immediate release (IR) methylphenidate (MPH). The clinical advantages offered by this novel compound go beyond ease of administration. By avoiding the peaks and valleys of serum levels associated with IR MPH, treatment with Concerta minimizes adverse effects at peaks and break through symptoms at valleys securing clinical coverage throughout the day, minimizing the risks of adverse effects from serum fluctuations that can occur with multiple dosing of the IR formulation of MPH. This unique pharmacokinetic and pharmacodynamic profile of Concerta is potentially particularly advantageous in the treatment of adults with ADHD because a) adults with ADHD tend to be forgetful; b) forgetfulness makes the self administration of treatment three times a day difficult; c) forgetfulness can lead to poor compliance and drop off of effects over time with its attendant detrimental effect on clinical control and quality of life. Subjects will be randomized by the pharmacy to CONCERTA or to continue MPH IR TID in a ratio of 4:1.

This study includes: 1) a six-week design to document the response rate 2) assessment of the impact of either MPH IR or Concerta on functional capacities 3) careful assessment of safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Male and female outpatients older than 18 and younger than 55 years of age.
3. If female, non-pregnant, non-nursing with a negative urine pregnancy test and using medically accepted means of birth control (abstinence, birth control pills, IUD, barrier devices, or progesterone rods stabilized for at least three months) while in this study.
4. Responders to methylphenidate IR on stable treatment (Stable treatment is defined as a score on the NIMH CGI improvement scale of much or very improved (compared to pre-treatment) from a period of 4 weeks on a stable dose of MPH IR TID).
5. Responders to methylphenidate IR on stable treatment who are satisfied with their treatment (satisfaction with treatment is defined as a score of 1 or 2 on the Treatment Satisfaction Rating scale from a period of 4 weeks on a stable dose of MPH IR TID).
6. Responders to methylphenidate IR on stable treatment who tolerate their treatment (toleration of treatment is defined as a score on the Tolerability Index of 0 or 1) from a period of 4 weeks on a stable dose of MPH IR TID).
7. Mild cases of asthma and allergy.
8. Acid reflux syndrome.
9. Hypercholesterolemia.
10. Subjects with a past history of tics but tic free for > 1 year.
11. Subjects with past history of depression, anxiety disorder (including OCD) without current disorder for > 6 months as ascertained through structured diagnostic interview and clinical exam.
12. Subjects treated for anxiety disorders (including OCD), and depression who are on a stable medication regimen for at least three months, and who have a disorder specific CGI-severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-anxiety rating scale below 15 (mild range) will be included in the study.
13. Subjects receiving non-MAOI antidepressants (e.g., SSRI's, venlafaxine), benzodiazepines, on a stable regimen for > 3 months for any of the conditions listed above.

Exclusion Criteria:

1. Diagnosis of, or family history of Tourette's syndrome, or Autism.
2. History of seizures.
3. Subjects with history of tics in the past year.
4. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence.
5. Any clinically unstable psychiatric conditions including the following: bipolar disorder, acute psychosis, acute panic, acute OCD, acute mania, acute suicidality, acute substance use disorders (alcohol or drugs), acute OCD, sociopathy, criminality or delinquency.
6. Subjects currently (within the past 4 weeks) receiving bupropion.
7. Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, opthalmic, or endocrine disease.
8. Clinically significant abnormal baseline laboratory values, which include the following:

   * Values larger than 20% above the upper range of the laboratory standard of a basic metabolic screen.
   * Exclusionary blood pressure parameters will include any values above 140 (systolic) and 90 (diastolic).
   * Exclusionary ECG parameters will include a QTC> 460msec, QRS>120 msec, and PR>200 msec. Any subject having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
9. Organic brain disorders.
10. Mental impairment as evidenced by an I.Q. <70 as determined by an abbreviated version of the Wechsler Adult Intelligence Scales (Wechsler Adult Intelligence Scales-Revised (WAIS-III) and the Wide Range Achievement Test (WRAT-III).
11. Pregnancy or lactation.
12. Glaucoma.
13. Non English speaking subjects will not be allowed into the study for the following reasons: a) the assessment instruments are not available and have not been adequately standardized in other languages; b) our clinical trials facility is located in Cambridge and not in the MGH main campus without the availability of translators; and c) even if such translation services were to be available, the assessments in the English language conducted by English speaking clinicians and raters with English speaking subjects is already extremely time consuming lasting many hours making it unfeasible, unrealistic, and of dubious clinical validity to conduct them with a translator with non English speaking subjects; d) psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: maintenance of symptom control when switched from TID IR MPH to Concerta administered once a day in the AM and to assess if this differs from 100%, the value one would expect if Concerta maintained efficacy in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States